CLINICAL TRIAL: NCT05064553
Title: ALTUS: Performance of a Multi- Target Hepatocellular Carcinoma (HCC) Test in Subjects With Increased Risk
Status: Active, not recruiting | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-01
Record Dates: First submitted 2021-09-21; First posted 2021-10-01 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-06

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer; Hepatitis B; Cirrhosis; Liver Cancer
Keywords: Blood Sample Collection; CT/MRI; Ultrasound; Combined Hepatocellular and Cholangiocarcinoma; HCC Surveillance
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Hepatitis B; Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be labeled with unique codes containing letters and numbers. Blood specimens may not be used in their entirety. Residual samples and their derivatives may be archived indefinitely for further analysis and future research. Specimens that are not processed, or specimens de-accessioned from the biorepository, will be destroyed with a record of removal and destruction maintained for seven years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ultrasound Surveillance Group: Subjects will undergo standard of care ultrasound surveillance imaging. Subjects with positive ultrasound are anticipated to have standard of care imaging follow-up with CT or MRI as well as other procedures as needed. Subjects with negative ultrasound will be sent for a study CT/MRI.
  Interventions: Device: Study CT/MRI Imaging; Device: Standard of Care CT/MRI Imaging; Diagnostic Test: Oncoguard™ Liver Test
- CT/MRI Surveillance Group: Subjects will undergo standard of care CT/MRI surveillance imaging.
  Interventions: Device: Standard of Care CT/MRI Imaging; Diagnostic Test: Oncoguard™ Liver Test

INTERVENTIONS:
Device: Study CT/MRI Imaging — Subjects with negative ultrasound will be sent for a study CT/MRI.
  Groups: Ultrasound Surveillance Group
Device: Standard of Care CT/MRI Imaging — Subjects with positive ultrasound are anticipated to have standard of care imaging follow-up as well as other procedures as needed.
Diagnostic Test: Oncoguard™ Liver Test — Subjects will have a blood sample collected for the Oncoguard™ Liver Test.

SUMMARY:
The primary objective is to assess overall sensitivity and specificity of Oncoguard™ Liver for hepatocellular cancer (HCC) detection in a surveillance population.

DETAILED DESCRIPTION:
The study will include participants aged 18 years and older who are at increased risk for HCC, including individuals with liver cirrhosis or non-cirrhotic individuals with chronic hepatitis B infection.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older.
2. Understand the study procedures, be able to provide written informed consent to participate in the study, and have authorization for release of data, including personal health data and images, to the study Investigator, Sponsor, and regulatory authorities.
3. Present for surveillance imaging due to increased risk for HCC, including either:

   1. Diagnosis of cirrhosis based on at least one of the following:

      * Histology from a liver biopsy.
      * Ultrasound, CT, or MRI showing a cirrhotic liver combined with portal hypertension (as evidenced by the presence of intra-abdominal varices, or recanalized umbilical vein, or ascites or splenomegaly or thrombocytopenia [defined as Platelet count < 150,000]). The imaging results must have been obtained within 5 years of study enrollment.
      * Liver stiffness ≥4.71 kilopascal (kPa) by Magnetic Resonance (MR) elastography or ≥12.1 kPa by vibration controlled transient elastography.
      * Presence of varices on endoscopy or imaging and presence of a chronic liver disease. Endoscopy or imaging results must have been obtained within 5 years of study enrollment.

      OR
   2. Non-cirrhotic subjects with chronic Hepatitis B Virus (HBV) infection (Hepatitis B surface antigen present for >6 months)

Exclusion Criteria:

1. Known cancer diagnosis (including active malignancy) within the past 5 years except for nonmelanoma skin cancer.
2. Chemotherapy and/or radiation therapy within 5 years prior to study enrollment.
3. Known Child-Pugh class C liver function at the time of enrollment, except for those on the waiting list for transplant.
4. Solid liver nodule >1 cm by ultrasound or elevated Alpha-fetoprotein (AFP) (>100 ng/mL) in 12 months preceding the qualifying surveillance imaging visit without subsequent documentation of HCC negative or LIRADS 1 (Liver Imaging Reporting and Data System) by diagnostic CT/MRI.
5. Females known to be pregnant at the time of enrollment.
6. Illness that the Investigator believes poses a significant risk of mortality during the study period, including but not limited to

   1. Congestive heart failure with ejection fraction <50%
   2. Chronic lung disease requiring supplemental oxygen.
   3. History of recent stroke.
7. Sustained virologic response (SVR) for Hepatitis C Virus (HCV) (undetectable HCV RNA 12 to 24 weeks after completion of antiviral therapy) for >10 years prior to enrollment.
8. Not able to have IV contrast for CT or MRI due to

   1. Allergy to IV contrast and unwilling or unable to receive IV contrast after pre-medication.
   2. Estimated glomerular filtration rate <35 mL/min and not on hemodialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects 18 years of age and older who are at an increased risk for HCC and for whom HCC surveillance is appropriate, including subjects with cirrhosis and non-cirrhotic subjects with Hepatitis B.
Sampling Method: Non-Probability Sample
Enrollment: 2990 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To demonstrate that Oncoguard™ Liver early-stage HCC sensitivity is non-inferior to that of ultrasound within a 5% margin | A maximum of 30 days from study or standard-of-care CT or MRI exam.
To demonstrate that Oncoguard™ Liver HCC specificity exceeds 82% | A maximum of 30 days from study or standard-of-care CT or MRI exam.

SECONDARY OUTCOMES:
To determine a point estimate and 95% confidence interval for Oncoguard™ Liver overall HCC sensitivity | A maximum of 30 days from study or standard-of-care CT or MRI exam.

CONTACTS AND LOCATIONS:
Overall Officials: Binu John, Principal Investigator — Miami VA Healthcare System
Locations (76):
- United States (76):
  - Arizona Health Research, Chandler, Arizona
  - Arizona Digestive Health - Sun City, Sun City, Arizona
  - Franco Felizarta, MD, Bakersfield, California
  - Gastroenterology & Liver Institute, Escondido, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Providence Facey Medical Foundation, Mission Hills, California
  - United Medical Doctors, Murrieta, California
  - VA Palo Alto Healthcare System, Palo Alto, California
  - Stanford University Medical Center, Palo Alto, California
  - California Liver Research Institute, Pasadena, California
  - Cadena Care Institute, Poway, California
  - Inland Empire Clinical Trials, Rialto, California
  - Research & Education, Inc, San Diego, California
  - San Jose Gastroenterology, San Jose, California
  - Rocky Mountain Gastroenterology, Littleton, Colorado
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - University of Florida Hepatology Research at CTRB, Gainesville, Florida
  - University of Florida - College of Medicine, Jacksonville, Florida
  - ENCORE Borland Groover Clinical Research, Jacksonville, Florida
  - Florida Research Institute, Lakewood, Florida
  - Miami VA Healthcare System, Miami, Florida
  - University of Miami, Miami, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Tampa General Hospital, Tampa Bay, Florida
  - Digestive Health Services, Downers Grove, Illinois
  - Illinois Gastroenterology Group, Glenview, Illinois
  - GI Alliance of Illinois - Gurnee, Gurnee, Illinois
  - Gastroenterology and Internal Medicine Specialists, Lake Barrington, Illinois
  - Avicenna Clinical Research, Oak Lawn, Illinois
  - NAVREF - Indiana Institute for Medical Research (IIMC), Indianapolis, Indiana
  - Indiana University, Indianapolis, Indiana
  - Indianapolis Gastroenterology Research Foundation, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Patient First Clinical Trials, Nottingham, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Southern Therapy and Advanced Research LLC (STAR), Jackson, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Brooklyn VA Medical Center, Brooklyn, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Manhattan Clinical Research, LLC, New York, New York
  - Digestive Health Partners, Asheville, North Carolina
  - Duke University Health Systems, Durham, North Carolina
  - VA North East Ohio Health Care System, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Great Lakes Medical Research - Susquehanna Research Group, Camp Hill, Pennsylvania
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Xiaoli MA MD, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Wilkes-Barre VA Medical Center, Wilkes-Barre, Pennsylvania
  - University Gastroenterology West River, Providence, Rhode Island
  - Ralph H Johnson VAMC, Charleston, South Carolina
  - Gastro One, Germantown, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Gastro Clinic, El Paso, Texas
  - Baylor - Saint Luke's Medical Center, Houston, Texas
  - Lubbock Digestive Disease Associates, Lubbock, Texas
  - Texas Digestive Disease Consultants - San Marcos, San Marcos, Texas
  - Tranquil Clinical Research, Webster, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - UVA Gastroenterology, Charlottesville, Virginia
  - Gastroenterology Associates, PC, Manassas, Virginia
  - Digestive & Liver Disease Specialists, Norfolk, Virginia
  - Bon Secours Liver Institute of Richmond, Richmond, Virginia
  - Richmond VA Medical Center, Richmond, Virginia
  - Washington Gastroenterology - Bellevue, Bellevue, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Velocity Clinical Research, Spokane, Washington
  - Washington Gastroenterology - Tacoma, Tacoma, Washington
  - UW Digestive Health Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include test, tables, figures, and appendices. The study protocol, statistical analysis plan (when applicable), informed consent form (when applicable), and the clinical study report (when applicable) will also be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available from 2 years and ending 4 years after publication.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/IEC approvals or waivers as applicable to conduct research.